CLINICAL TRIAL: NCT02750722
Title: Acute Effects of Combined Exercise and Oscillatory Positive Expiratory Pressure Therapy on Sputum Properties and Lung Diffusion Capacity in Cystic Fibrosis: a Randomized Crossover Trial
Brief Title: Exercise and Oscillatory Positive Expiratory Pressure Therapy in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-00153
Record Dates: First submitted 2016-04-12; First posted 2016-04-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Cystic Fibrosis
Keywords: Exercise; Lung diffusion capacity; Sputum viscoelasticity; Lung disease
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity; Lung Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cycling in combination with Flutter® therapy (Experimental): Participants perform 30 minutes of moderately intense cycling exercise in 4-min intervals at 75% of their maximal heart rate and interspersed with 2-min resting periods during which 6-8 breathing maneuvers are performed with the Flutter®.
  Interventions: Device: Flutter®
- Cycling without Flutter® therapy (Active Comparator): Participants perform 30 minutes of continuous moderately intense cycling exercise at 75% of their maximal heart rate without additional Flutter® breathing maneuvers.
  Interventions: Device: No Flutter®

INTERVENTIONS:
Device: Flutter® — Acute exercise with Flutter® breathing therapy.
  Arms: Cycling in combination with Flutter® therapy
Device: No Flutter® — Acute exercise without Flutter® breathing therapy.
  Arms: Cycling without Flutter® therapy

SUMMARY:
The investigators aim to compare a single bout of moderately intense cycling exercise incorporating Flutter® breathing maneuvers with a single bout of moderately intense cycling exercise alone on sputum viscoelasticity (primary endpoint) and the diffusion capacity of the lungs in adult patients with cystic fibrosis.

The investigators further aim to analyze the short-term variability of resting diffusion capacity of carbon monoxide (DLCO) and nitric oxide (DLNO) in patients with cystic fibrosis.

DETAILED DESCRIPTION:
Regular airway clearance is an integral component of cystic fibrosis care and of critical importance to lung health. Exercise and standardized chest physiotherapy are accepted airway clearance techniques in cystic fibrosis. Different airway clearance techniques are available, but there is no evidence that one technique or a combination is superior. Oscillatory positive expiratory pressure with the Flutter® is a widely used airway clearance technique in the European countries and has been shown to favourably alter sputum viscoelasticity in cystic fibrosis.

This randomized crossover study is designed to assess the acute effects of combined cycling exercise and Flutter® therapy on sputum viscoelasticity (primary outcome measure) and gas diffusion in adults with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF based on either two CF-causing mutations and/or a sweat chloride concentration during two tests of > 60 mmol/l
* Patients that are able to provide sputum samples
* Adult age ≥ 18 years

Exclusion Criteria:

* Unstable condition affecting participation in the exercise experiments (i.e., major hemoptysis or pneumothorax within the last 3 months, acute exacerbation and iv-antibiotics during the last 4 weeks, unstable allergic bronchopulmonary aspergillosis, listed for lung transplantation, major musculoskeletal injuries such as fractures or sprains during the last 2 months, others according to the impression of the doctor)
* Cardiac arrhythmias with exercise
* Requiring additional oxygen with exercise
* Colonization with Burkholderia cenocepacia
* Status post lung transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-01-19 (Actual); Study Completion 2017-01-19 (Actual)

PRIMARY OUTCOMES:
Change in sputum viscoelasticity (G*) over a broad frequency range (1-100 rad.s-1) | Baseline - immediately post exercise - 45min post exercise
  Sputum viscoelasticity measured by stress/strain controlled rheometer (Anton Paar, MCR 301/MCR 501).

SECONDARY OUTCOMES:
Change in shear viscosity (η) | Baseline - immediately post exercise - 45min post exercise
  Shear viscosity measured by stress/strain controlled rheometer (Anton Paar, MCR 301/MCR 501).
Change in sputum spinnability (mm) | Baseline - immediately post exercise - 45min post exercise
  Measured with a Capillary Breakup Extensional Rheometer (CaBER).
Change in sputum solids content (%) | Baseline - immediately post exercise - 45min post exercise
  Sputum weight of a 50 μL aliquot before and after lyophilization to dryness using a freeze dryer.
Change in lung diffusion capacity for nitric oxide (DLNO) | Baseline - immediately post exercise - 45min post exercise
  Single-breath measurements with MasterScreenTM PFT system
Change in lung diffusion capacity for carbon monoxide (DLCO) | Baseline - immediately post exercise - 45min post exercise
  Single-breath measurements with MasterScreenTM PFT system
Change in DLNO/DLCO ratio | Baseline - immediately post exercise - 45min post exercise
  Single-breath measurements with MasterScreenTM PFT system
Change in alveolar volume | Baseline - immediately post exercise - 45min post exercise
  Single-breath measurements with MasterScreenTM PFT system
Change in pulmonary capillary blood volume | Baseline - immediately post exercise - 45min post exercise
  Single-breath measurements with MasterScreenTM PFT system
Change in pulmonary membrane diffusion capacity | Baseline - immediately post exercise - 45min post exercise
  Single-breath measurements with MasterScreenTM PFT system
Change in ease of sputum expectoration (cm) | Baseline - immediately post exercise - 45min post exercise
  Assessed by a visual analogue scale (0-10)
Change in oxygen saturation (%) | Baseline - immediately post exercise - 45min post exercise
  Measured by pulse oximetry.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Radtke, PhD, Principal Investigator — University of Zurich
Locations (3):
- Switzerland (3):
  - University of Zurich, Zurich, Canton of Zurich
  - University Hospital Zurich, Zurich, Canton of Zurich
  - ETH Zurich, Zurich, Canton of Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Radtke T, Boni L, Bohnacker P, Maggi-Beba M, Fischer P, Kriemler S, Benden C, Dressel H. Acute effects of combined exercise and oscillatory positive expiratory pressure therapy on sputum properties and lung diffusing capacity in cystic fibrosis: a randomized, controlled, crossover trial. BMC Pulm Med. 2018 Jun 14;18(1):99. doi: 10.1186/s12890-018-0661-1. PMID 29898704